CLINICAL TRIAL: NCT04933682
Title: A Phase 1 Two-Part Study to Evaluate the Potential Drug Interactions Between ALXN2050 and Fluconazole, and Between ALXN2050 and Rifampin in Healthy Adult Participants
Brief Title: Drug Interaction Study of ALXN2050 With Fluconazole and Rifampin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-105
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: ALXN2050; Fluconazole; Rifampin; Drug-Drug Interaction
MeSH Terms: interventions — rhoA GTP-Binding Protein; Fluconazole; Rifampin

STUDY DESIGN:
Intervention Model Description: This will be a 2-part, open-label, fixed-sequence study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: ALXN2050 plus Fluconazole (Experimental): Period 1: Participants will receive a single dose of ALXN2050 alone and in the presence of multiple doses of fluconazole.
  Period 2: Participants will receive multiple doses of ALXN2050 alone and in the presence of multiple doses of fluconazole.
  Scheduled pharmacokinetics (PK) blood samples for both ALXN2050 and fluconazole will be collected, with a washout period of at least 14 days between the last dose of fluconazole in Period 1 and the first dose of ALXN2050 in Period 2.
  Interventions: Drug: ALXN2050; Drug: Fluconazole
- Part 2: ALXN2050 plus Rifampin (Experimental): Participants will receive a single dose of ALXN2050 alone and in the presence of both single and multiple doses of rifampin.
  Scheduled PK blood samples for both ALXN2050 and rifampin will be collected.
  Interventions: Drug: ALXN2050; Drug: Rifampin

INTERVENTIONS:
Drug: ALXN2050 — Oral tablet.
  Other Names: ACH-0145228 (formerly)
Drug: Fluconazole — Oral tablet.
  Arms: Part 1: ALXN2050 plus Fluconazole
Drug: Rifampin — Oral capsule.
  Arms: Part 2: ALXN2050 plus Rifampin

SUMMARY:
This is a 2-part, open label, fixed-sequence study to evaluate the potential drug interaction between ALXN2050 and fluconazole (Part 1), and between ALXN2050 and rifampin (Part 2) in healthy adult participants. Part 1 will be a 2-period, fixed-sequence study. Part 2 will be a single-period, fixed-sequence study.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically healthy with no clinically significant or relevant abnormalities as determined by medical history, physical or neurological examination, vital signs, 12-lead electrocardiogram, screening clinical laboratory profiles.
* Body mass index within the range 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at Screening.

Key Exclusion Criteria:

* History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* History of significant multiple and/or severe allergies.
* Any previous procedure that could alter absorption or excretion of orally administered drugs.
* Participation in another investigational drug or investigational device study within 5 half-lives (if known) or 30 days prior to the first dose of study intervention, whichever is longer.
* Body temperature ≥ 38.0°Celsius, at Screening or prior to the first dose of study intervention.
* History of drug or alcohol abuse within 2 years prior to the first dose of study intervention or positive drugs-of-abuse or alcohol screen at Screening or Day -1; current tobacco/nicotine user or smoker or a positive cotinine test at Screening.
* Donation of whole blood from 3 months prior to the first dose of study intervention, or of plasma from 30 days prior to the first dose of study intervention; receipt of blood products within 6 months prior to the first dose of study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Part 1: Area Under The Concentration-time Curve From Time 0 To Infinity (AUC0-inf) For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Fluconazole | Up to 72 hours postdose
Part 1: Maximum Observed Concentration (Cmax) For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Fluconazole | Up to 72 hours postdose
Part 1: Time To Maximum Plasma Concentration (Tmax) For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Fluconazole | Up to 72 hours postdose
Part 1: Area Under The Concentration-time Curve From Time 0 To The 12-hour Point (AUC0-12) For Multiple Doses Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Fluconazole | Up to 72 hours postdose
Part 1: Cmax For Multiple Doses Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Fluconazole | Up to 72 hours postdose
Part 1: Tmax For Multiple Doses Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Fluconazole | Up to 72 hours postdose
Part 2: AUC0-inf For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed With A Single Dose Of Rifampin | Up to 72 hours postdose
Part 2: Cmax For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed With A Single Dose Of Rifampin | Up to 72 hours postdose
Part 2: Tmax For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed With A Single Dose Of Rifampin | Up to 72 hours postdose
Part 2: AUC0-inf For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Rifampin | Up to 72 hours postdose
Part 2: Cmax For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Rifampin | Up to 72 hours postdose
Part 2: Tmax For A Single Dose Of ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Rifampin | Up to 72 hours postdose

SECONDARY OUTCOMES:
Part 1: Area Under The Concentration-time Curve From Time Zero To The 4-hour Time Point (AUC0-4) For ALXN2050 When Dosed In The Morning Versus In The Evening | Up to 12 hours postdose
Participants Experiencing Treatment-emergent Adverse Events | Up to 40 days postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No